CLINICAL TRIAL: NCT02450903
Title: A Phase II, Multi-center, Open-label, Single-Arm Study to Evaluate the Efficacy and Safety of Oral LDK378 Treatment for Patients With ALK-Positive Non-Small Cell Lung Cancer Previously Treated With Alectinib
Brief Title: LDK378 in Patients With ALK Positive NSCLC Previously Treated With Alectinib.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A1201
Record Dates: First submitted 2015-05-08; First posted 2015-05-21 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-01

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; NSCLC; ALK; LDK378; alectinib; Non-small cell lung carcinoma (NSCLC); lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; Non small cell lung cancer; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDK378 (Ceritinib) (Experimental): Participants who received LDK378 750mg once daily on a 28 day cycle.
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — Oral LDK378 750mg once daily
  Other Names: Oral LDK378 750mg once daily

SUMMARY:
This was a single-arm, open-label, multicenter, phase II study to evaluate the efficacy and safety of the ALK inhibitor LDK378 when used as single agent in patients with ALK-rearranged stage IIIB or IV NSCLC previously treated with alectinib. Treatment with LDK378 750 mg qd continued until the patient experienced disease progression as determined by the investigator according to RECIST 1.1, unacceptable toxicity that precluded further treatment, pregnancy, start of a new anticancer therapy, discontinued treatment at the discretion of the patient or investigator, lost to follow-up, death, or study was terminated by Sponsor.

DETAILED DESCRIPTION:
Study completed as per protocol. 'Switched to commercial drug' implies that after the primary and secondary objectives were achieved, one patient continued the study treatment as they did not meet the progression disease or AE to be discontinued from the treatment. But after the regulatory approval, Novartis decided to close the study, the 1 patient switched to commercially available drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Stage IIIb or IV NSCLC that carries an ALK rearrangement as determined locally by Vysis ALK Break Apart FISH Probe Kit (Abbott Molecular Inc.) test.
* Patients must have NSCLC that has progressed at study enrollment.
* Patients must have received previous treatment with alectinib for treatment of locally advanced or metastatic NSCLC. Prior therapy with crizotinib as ALK inhibitor therapy in addition to alectinib is allowed. Alectinib doesn't need to be the last therapy prior to study enrollment. No particular sequence of prior alectinib and crizotinib is required for enrollment.
* Patients must be chemotherapy-naïve or have received only one line of prior cytotoxic chemotherapy.
* Age 18 years or older at the time of informed consent.

Key Exclusion Criteria:

* Patients with known hypersensitivity to any of the excipients of LDK378.
* Prior therapy with other ALK inhibitor investigational agents except crizotinib and alectinib.
* Prior systemic anti-cancer (including investigational) therapy aside from alectinib, crizotinib and one regimen of previous cytotoxic chemotherapy for locally advanced or metastatic NSCLC.
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Patient with history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis.
* Patients with history of carcinomatous meningitis.
* Patient with a concurrent malignancy or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years.
* Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sakyo Ku, Kyoto
  - Novartis Investigative Site, Natori-shi, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hida T, Seto T, Horinouchi H, Maemondo M, Takeda M, Hotta K, Hirai F, Kim YH, Matsumoto S, Ito M, Ayukawa K, Tokushige K, Yonemura M, Mitsudomi T, Nishio M. Phase II study of ceritinib in alectinib-pretreated patients with anaplastic lymphoma kinase-rearranged metastatic non-small-cell lung cancer in Japan: ASCEND-9. Cancer Sci. 2018 Sep;109(9):2863-2872. doi: 10.1111/cas.13721. Epub 2018 Jul 25. PMID 29959809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 20 patients were planned to be enrolled.
Pre-assignment Details: A total of 20 patients were enrolled and treated with ceritinib.
Period: Overall Study
Arm/Group | LDK378 (Ceritinib)
Started | 20
Entered Post-treatment Effic. f/u Phase (Discontinued from treatment phase) | 4
Entered Survival Follow-up Phase (Discontinued from treatment phase) | 15
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 3
Not completed — Progressive disease | 15
Not completed — Switched to commercial drug | 1
Not completed — Subject/guardian decision | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib. Safety Set in this study is identical to FAS.
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (15.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 19
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) to LDK378 by Investigator Assessment
Description: ORR, defined as the percentage of participants with a best overall confirmed response of complete response (CR) or partial response (PR) in the whole body as assessed per RECIST 1.1 by the investigator. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Until disease progression or unacceptable toxicity occurs, or patient withdrawal up to 798 days
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 20
Percentage of participants | 25.0 [8.7 to 49.1]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR, calculated as the percentage of participants with best overall response of CR, PR, or stable disease (SD) evaluated by investigator per RECIST 1.1; CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD); PD: taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: 6 cycles of 28 days up to 798 days
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 20
Percentage of participants | 70.0 [45.7 to 88.1]

3. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR, calculated as the time from first dose of LDK378 to first documented response (CR or PR) evaluated by investigator per RECIST 1.1 for participants with confirmed PR or CR.
Time Frame: 6 cycles of 28 days up to 798 days
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib - participants with confirmed PR or CR.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 5
Months | 1.8 (0.0818)

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR, calculated as the time from the date of the first documented response (CR or PR) to the first documented disease progression evaluated by investigator per RECIST 1.1 or death due to any cause
Time Frame: 6 cycles of 28 days up to 798 days
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 5
Months | 6.3 [3.5 to 9.2]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, calculated as the time from first dose of LDK378 to date of first documented disease progression evaluated by investigator per RECIST 1.1 or date of death due to any cause
Time Frame: 6 cycles of 28 days up to 798 days
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 20
Months | 3.7 [1.9 to 5.3]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start date of study drug to the date of death due to any cause.
Time Frame: 6 cycles of 28 days up to 798 days
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 20
Months | 17.3 [9.1 to NA] — N/A= not enough number of events to calculate the upper limit of the confidence interval.

7. Secondary Outcome: Overall Intracranial Response Rate (OIRR)
Description: OIRR, calculated as the percentage of participants with a best overall confirmed response of CR or PR in the brain assessments for participants having measurable brain metastases at baseline
Time Frame: 6 cycles of 28 days up to 798 days
Population: Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib - participants with measurable brain disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 2
Percentage of participants | 0.0 [0.0 to 84.2]

8. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 24 months (treatment duration ranged from 0.4 to to 23.0 months). Deaths post treatment survival follow up were collected after the on treatment period, up to 33 months. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: approx. 24 months, approx. 33 months
Population: Clinical Database Population: all treated patients and patients who died during screening
Measure: Number; unit: Participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 20
Participants
  Total Deaths | 12
  Deaths on-treatment | 0
  Deaths post-treatment survival follow-up | 12

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 24 months (treatment duration ranged from 0.4 to to 23.0 months).
Description: AE: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | LDK378 (Ceritinib)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 (Ceritinib) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1
Hepatobiliary disease (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 (Ceritinib) (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 8
Amylase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 2
Blood creatinine increased (Investigations) | 9
Electrocardiogram QT prolonged (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 2
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02450903/SAP_000.pdf
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT02450903/Prot_001.pdf